CLINICAL TRIAL: NCT06931509
Title: Study of the Integration and Interactions Between Visual and Proprioceptive Feedbacks in Hemiplegic Patients
Brief Title: Integration and Interactions Between Visual and Proprioceptive Feedbacks
Acronym: OptiVis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24CH167; 2024-A02163-44 (Other: ANSM)
Record Dates: First submitted 2025-03-25; First posted 2025-04-17 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Hemiparetic Stroke
Keywords: Computerize mirror; Vibration; Upper limb rehabilitation; Stroke; hemiplegic
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computerized mirror therapy (IVS3) + Tendon vibration (Vibramoov) (Experimental): During these sessions, they will perform a wrist extension task 30 times, under four different rehabilitation conditions (in randomized order), with pauses between conditions:
  * Movement without feedback
  * Movement with visual feedback
  * Movement and vibratory feedback
  * Movement with combined visual and vibratory feedback. Visual and vibratory feedback is provided using the IVS3 and Vibramoov Physio devices.
  Interventions: Device: Computerized mirror therapy (IVS3) + Tendon vibration (Vibramoov)

INTERVENTIONS:
Device: Computerized mirror therapy (IVS3) + Tendon vibration (Vibramoov) — Visit 1 : Followed by 30 movements of Paretic arm wrist extension with 4 randomized experimental conditions (Vision alone, Vibration alone, Vision + Vibration, No feedback), with EEG monitoring. Measurement of movement perception feeling for each condition.
  Visit 2 : 30 movements of Paretic arm wrist extension with 4 randomized experimental conditions (Vision alone, Vibration alone, Vision + Vibration, No feedback), with EEG monitoring. Measurement of movement perception feeling for each condition.

SUMMARY:
Mental imagery is a rehabilitation technique for stroke patients, involving the mental representation of movement. Recent technical advancements have enabled the use of visual, proprioceptive, and mixed feedback to enhance motor stimulation. Currently, all post-stroke patients receive these techniques indiscriminately. This study aims to demonstrate differences in the integration of visual and proprioceptive feedback in stroke patients and understand the determinants based on the affected brain area.

Patients with motor disabilities will perform motor imagery tasks with various feedback types while their cortical activity is recorded using EEG. EEG data for each type of feedback will be correlated with the lesion area in order to better understand the ongoing mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic subjects : Male or female, aged 18 to 80 years, first ischemic or hemorrhagic stroke, having signed the written consent and affiliated or entitled to a social security scheme

Exclusion Criteria:

* Severe cognitive impairment, severe Aphasia or severe neglect that impair ability to understand instructions or to execute tasks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
EEG beta desynchronization | Day 1
  Differences in the EEG beta desynchronization over motor-cortex across the types of feedbacks.

SECONDARY OUTCOMES:
Alpha Band | Day 1
  Alpha Band desynchronization over motor cortex
Occipital alpha band | Day 1
  Occipital alpha band modulations
Beta rebound | Day 1
  Beta rebound (Event related synchronization)
Parietal beta-band | Day 1
  Parietal beta-band desynchronization
Perception of movements | Day 1
  The intensity of the perception of movements using a visual analogue scale and the objective measurement of perceived movement angle reproduced by the healthy hand's and Visual analogic scale

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Adham, Md, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France, France

IPD SHARING:
Plan to Share IPD: Undecided
The study is monocentric